CLINICAL TRIAL: NCT01470495
Title: Radiofrequency Ablation Plus Sorafenib Administration in Early Recurrent Hepatocellular Carcinoma: a Prospective Multicenter Cohort Trial (Repeat) Tumors for BCLC B Stage HCC Undergone Curative Hepatectomy
Brief Title: Combined Treatment of RFA and Sorafenib on Recurrent HCC
Acronym: REPEAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Collaborators: Hunan Province Tumor Hospital (Other); Tang-Du Hospital (Other); Xijing Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Anhui Provincial Hospital (Other Government); Xiangya Hospital of Central South University (Other); Xinqiao Hospital of Chongqing (Other); Xinjiang Tumor Hospital (Unknown); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Henan Cancer Hospital (Other Government); People's Hospital of Sichuan (Unknown); Huaxi Hospital (Other)
Responsible Party: Principal Investigator, feng xiaobin, Institute of hepatobiliary surgery,southwest hospital, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: swhb005
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: HCC; Radiofrequency Ablation; Sorafenib
MeSH Terms: interventions — Radiofrequency Ablation; Sorafenib

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA+Sorafenib (Experimental): to treat recurrent HCC both with RFA and Sorafenib
  Interventions: Other: RFA + Sorafenib
- RFA group (Active Comparator): To treat recurrent HCC with RFA
  Interventions: Other: RFA

INTERVENTIONS:
Other: RFA + Sorafenib — combined RFA and Sorafenib to treat recurrent HCC
  Arms: RFA+Sorafenib
Other: RFA — treat Recurrent HCC with RFA
  Arms: RFA group

SUMMARY:
RFA is a routaine treatment of recurrent HCC. Recently Sorafenib was reported to be a promising drug to treat late stage HCC. But few studies were related with its effectiveness on recurrent HCC. So the investigators hypothesized that combined RFA and Sorafenib might reduce the frequency of recurrence and improve the overall survival and disease free survial.

ELIGIBILITY:
Inclusion Criteria:

* recurrent HCC after curative resection
* without gender restriction
* age between 18 to 75 years
* The liver function showed no worse than Child-Pugh B
* tumor nodes were less than 5cm and no more than 3 nodules

Exclusion Criteria:

* Pregnancy patients
* With extrahepatic tumor or lymphnode metastasis
* Tumor invasion or thrombosis in portal vein,hepatic vein or inferior vena cava

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
time interval between new lessions emerging after the first HCC recurrence | 3 year

SECONDARY OUTCOMES:
3-year overrall survival | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Kuansheng Ma, MD,Ph.D, Principal Investigator — Southwest Hopstial
Locations (1):
- Institute of hepatobiliary surgery,southwest hospital, Chongqing, Chongqing Municipality, China